CLINICAL TRIAL: NCT07100938
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of BGB-45035 Versus Placebo in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: A Study Investigating the Efficacy and Safety of BGB-45035 Versus Placebo in Adults With Moderate to Severe Active Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-45035-201
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Interleukin-1 Receptor-Associated Kinase 4 (IRAK4) Degrader
MeSH Terms: conditions — Arthritis, Rheumatoid; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BGB-45035 (Experimental): Participants will receive BGB-45035 orally for up to 12 weeks
  Interventions: Drug: BGB-45035
- Placebo (Placebo Comparator): Participants will receive placebo orally for up to 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGB-45035 — Administered orally
  Arms: BGB-45035
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
This study aims to evaluate the efficacy of BGB-45035 in adults with moderate to severe active rheumatoid arthritis (RA) who have had an inadequate response to conventional synthetic disease-modifying antirheumatic drugs (csDMARDs) or biologic disease-modifying antirheumatic drugs (bDMARDs)/targeted synthetic disease-modifying antirheumatic drugs (tsDMARDs).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis (RA) based on American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria for at least 3 months prior to screening
* Demonstrated an inadequate response to, or loss of response or intolerance to at least 1 conventional synthetic disease-modifying antirheumatic drug (csDMARD) (Hydroxychloroquine, methotrexate [MTX], leflunomide, or sulfasalazine) or 1 biologic disease-modifying antirheumatic drug (bDMARD)/targeted synthetic disease-modifying antirheumatic drug (tsDMARD) treatment
* Must be on stable dose of one of the following permitted therapies for ≥ 4 weeks prior to screening and during the study: methotrexate between 7.5 mg to 25 mg/week, hydroxychloroquine up to 400 mg/day, leflunomide up to 20 mg/day, or sulfasalazine between 1000 mg/day to 3000 mg/day

Exclusion Criteria:

* Class IV RA based on American College of Rheumatology revised criteria for classification of functional status in rheumatoid arthritis
* Patients with a history of cancer in the last 5 years before the Screening Visit, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin
* Have failed more than 2 b/tsDMARDs (eg, excluded if have failed 2 bDMARDs and 1 tsDMARD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Disease Activity Score - C-reactive protein (DAS28-CRP) at Week 12 | Baseline and Week 12
  The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), high-sensitivity C-reactive protein (hsCRP in mg/L), and Patient's Global Assessment of Arthritis Pain (measured on a Visual Analog Scale [VAS] from 0 [no pain] to 100 [worst possible pain]). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity. A score greater than 5.1 indicates high disease activity, a score between 3.2 and 5.1 indicates moderate disease activity, a score between 2.6 and 3.2 indicates low disease activity, and a score less than 2.6 indicates the participant is in remission.

SECONDARY OUTCOMES:
Percentage of participants with a 20% improvement in American College of Rheumatology Criteria (ACR20) | Baseline and Week 12
  The ACR20 is defined as at least 20% improvement in the ACR core set values as defined below. Participants must meet 3 conditions for improvement from Baseline:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Percentage of participants with a 50% improvement in American College of Rheumatology Criteria (ACR50) | Baseline and Week 12
  The ACR50 is defined as at least 50% improvement in the ACR core set values as defined below. Participants must meet 3 conditions for improvement from Baseline:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Percentage of participants with a 70% improvement in American College of Rheumatology Criteria (ACR70) | Baseline and Week 12
  The ACR70 is defined as at least 70% improvement in the ACR core set values as defined below. Participants must meet 3 conditions for improvement from Baseline:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Change from Baseline in Tender Joint Count 68 (TJC 68) | Baseline up to Week 12
  The TJC 68 is an assessment of tenderness or pain in 68 joints. Sixty-eight joints will be assessed for tenderness/pain by an independent, blinded assessor. The response to pressure/motion on each joint is assessed using the following scale: Present/Absent/Not Done/Not Applicable. A lower score indicates there is less pain or tenderness present, while a higher score indicates more pain or tenderness is present.
Change from baseline in Swollen Joint Count 66 (SJC 66) | Baseline up to Week 12
  The SJC 66 is an assessment of swelling in 66 joints. Sixty-six joints will be assessed for swelling by an independent, blinded assessor. The swelling present in each joint is assessed using the following scale: Present/Absent/Not Done/Not Applicable. A lower score indicates there is less swelling present, while a higher score indicates more swelling is present.
Change from baseline in physician's global assessment of disease activity (PhGADA_VAS) | Baseline up to Week 12
  The PhGADA_VAS is a single item that asks the physician to assess the participant's current disease activity on a 0- to 100-mm visual analog scale (VAS), with anchors of 0 = "no disease activity" and 100 = "extremely active disease."
Change from baseline in Simplified Disease Activity Index (SDAI) score | Baseline up to Week 12
  The simplified disease activity index (SDAI) is a composite measure that sums the total number of:
  * 28 tender joint counts,
  * 28 swollen joint counts,
  * Patient's Global Assessment of Disease Activity measured on a VAS from 0 to 10 where 0= lowest disease activity and 10 = highest;
  * Physician's Global Assessment of Disease Activity measured on a VAS from 0 to 10, where 0 = lowest disease activity and 10 = highest, and
  * C-reactive protein (CRP) in mg/dL. The SDAI score ranges from 0 to approximately 86 where lower scores indicate less disease activity.
Change from baseline in Clinical Disease Activity Index (CDAI) score | Baseline up to Week 12
  The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the:
  * 28 tender joint count (TJC),
  * 28 swollen joint count (SJC),
  * Patient's Global Assessment of Disease Activity measured on a VAS from 0 to 10 where 0 = lowest disease activity and 10 = highest;
  * Physician's Global Assessment of Disease Activity (measured on a VAS from 0 to 10 where 0 = lowest disease activity and 10 = highest).
  The CDAI score ranges from 0 to 76 where lower scores indicate less disease activity.
Change from baseline of participant's global assessment of disease activity (PaGADA_VAS) | Baseline up to Week 12
  The PaGADA_VAS is a single item that asks the patient to rate the current severity of their disease activity on a 0- to 100-mm VAS, with anchors of 0 = "no disease activity" and 100 = "extremely active disease."
Change from baseline of Participant's global assessment of arthritis pain (VAS) | Baseline up to Week 12
  The Participants's global assessment of arthritis pain (VAS) is a single item that asks the patient to rate the current severity of their pain in relation to their RA on a 0- to 100-mm VAS, with anchors of "no pain" and "worst possible pain."
Change from baseline of Participant's assessment of physical function as measured by the Health Assessment Questionnaire - Disability Index (HAQ-DI) | Baseline up to Week 12
  The HAQ-DI is a patient-reported questionnaire that is commonly used in RA to measure disease-associated disability (assessment of physical function). Participants answer 24 questions using a scale from 0 to 3 to score difficulty when performing daily activities over the past week (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). Scores on each task are averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three represents very severe, high-dependency disability.
Number of participants with adverse events (AEs) | Up to approximately 4 months
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including findings from laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (26):
- China (26):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Chenzhou No Peoples Hospital, Chenzhou, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Northern Jiangsu Peoples Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Pingxiang Peoples Hospital, Pingxiang, Jiangxi
  - Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical Colleg, Nanchong, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/